CLINICAL TRIAL: NCT05937087
Title: Developing Community Partnerships Through Research to Define Community Well-Being From a Diné-centered Perspective With Three (Diné) Navajo Communities in New Mexico
Brief Title: Developing Community Partnerships Through Research to Define Community Well-Being With Three (Diné) Navajo Communities
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Vincent Robert Werito, Associate Professor, University of New Mexico
Other Study IDs: University of New Mexico
Record Dates: First submitted 2023-05-31; First posted 2023-07-10 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Behavior, Health; Mental Health Wellness 1; Community
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TOC community advisory research team: Participants were given a pre-and post community engagement survey.
  Interventions: Other: Community engaged research

INTERVENTIONS:
Other: Community engaged research — The university is working with Navajo communities to conduct an intervention study integrating community based participatory research using an Indigenous research paradigm. The innovative proposed project uses two approaches to build a research partnership to create capacity in the community for community-engaged multilevel behavioral and mental health research. Members from the three Navajo communities have never previously been involved in health research focused on wellbeing. Integrating CBPR with DCSR methodology becomes a powerful innovative intervention as the: 1) the community is driving the research to identify culture-based solutions for health related disparities; 2) the community is provided opportunities through research to center their perspectives and understandings about behavioral and mental health interventions; and 3) the community draws upon their collective community Indigenous knowledge.

SUMMARY:
This community engaged research pilot project begins a process of engaging Navajo community members from the communities of Counselor, Ojo Encino, and Torreon chapters in northwest New Mexico in critical dialogue and praxis to address longstanding health disparities. The research design is based on a Tribal Crit theoretical framework that aims to explore the perspectives of community members' understandings of wellbeing from a Diné centered paradigm using a community based participatory research approach integrated with a Diné-centered scientific research methodology. The proposed aims include using the Diné conceptualization of K'é (kinship) to define community wellbeing with future plans to build upon this knowledge by developing a community profile survey for obtaining baseline community health information that can be used to inform future research studies. A long-term goal of this mixed-method, community-based participatory research (CBPR) study is to create a community-university research partnership in an Indigenous context by establishing a multi-dimensional, Diné-centered research infrastructure with the capacity to improve mental/behavioral health outcomes and reduce health disparities. The creation of this infrastructure is a critical first step that will make it possible to use health research to positively transform the health landscape in Indigenous communities

DETAILED DESCRIPTION:
Specific Aims. Indigenous communities experience alarmingly high rates of depression, drug and alcohol dependency, school dropout, and suicide. For example, Indigenous youth suicide rates are at crisis levels. Unfortunately, research methods used to address these critical issues have often failed to provide sufficient understanding of the complex dynamics underpinning these challenges in Indigenous contexts. As a result, mental/behavioral health interventions have been largely unsuccessful, Indigenous health disparities have actually increased, and complex culture-based relationships that influence health outcomes are under conceptualized. Solutions to this health disparity dilemma require a new research paradigm. Past preliminary work in Indigenous communities in New Mexico (NM) has been illuminating in this respect which showed that a lack of wellbeing at individual, family, and community levels is associated with traumatic past experiences, a decline in Indigenous cultural practices, and decreasing use of the Indigenous language. And, in communities where the investigators worked, they were told that researchers have failed to involve community members or include community perspectives in the design or implementation of research and health interventions. Further, this preliminary work found that Indigenous community members associated the rise of 'fracking' activities on their lands by energy companies to negative behavioral/mental health outcomes that has implications for defining wellbeing from a Diné-centered perspective using a community driven research approach. This proposed mixed-method, community-based participatory research (CBPR) study builds on our previous work to develop a Diné-Centered Scientific Research (DCSR) methodology in three Navajo (Diné) communities in northwestern NM. The goal of this study is to create a community-university research partnership in an Indigenous context by establishing a multi-dimensional, Diné-centered research infrastructure with the capacity to improve mental/behavioral health outcomes and reduce disparities. The creation of this infrastructure is a critical first step that will make it possible to use health research to positively transform the health landscape in Indigenous communities.

Aim # 1. To create a community-driven understanding of the concept of research, research methods, and research protocols using CBPR and DCSR to develop a unique Diné multi-level behavioral health framework. Hypothesis: Creating a community-driven understanding of the concept of research, including purpose, ownership of data, methods, protocols, and research design will increase the ability of community members to understand what research means to them personally and as a community, decrease mistrust that often characterizes attempts to conduct research in such contexts, and to be clear on the implications of participating in research. Questions: a) What is the community-based concept of research that is articulated? b) How does existing community capacity enhance reflection on desired partnership values and strategies and how does this change in the process? c) How did creation of the partnership impact community trust? d) Did creation of the partnership decrease anxiety regarding community research? e). What collaboration factors are achieved/not achieved? Aim # 2. To enable the Diné culture-based concept of k'é (relationships) to evoke wellbeing that will be enacted as a culturally relevant framework for multilevel mental and behavioral health interventions. Hypothesis: Integrating a CBPR framework with a DCSR methodology will enable the Diné concept of K'é to empower our community partners to develop culturally based interventions to address community-identified health priorities. Questions: a) In what ways are the core cultural values of the community mobilized to address health disparities? b) What is the community-defined understanding of wellbeing? c) How can K'é, as a cultural strengths model, be used to facilitate community dialogue and praxis for transformative healing? d) How does K'é influence the way that local elders, traditional practitioners, and/or other community members are involved in the design and outcomes of behavioral and mental health interventions?

SIGNIFICANCE Devastating Mental and Behavioral Health Disparities in Indigenous Communities. Indigenous communities experience alarmingly high rates of depression, drug and alcohol dependency, and suicide. Indigenous youth suicide rates are at crisis levels. In a preliminary study, the investigators found that Navajo community members associated the rise of 'fracking' activities on their lands by energy companies to negative behavioral and mental health outcomes . However, mental/behavioral health interventions that have been designed for implementation in tribal settings using Western models have been largely unsuccessful, complex relationships that influence health outcomes are under conceptualized, and Indigenous health disparities have actually increased. Solutions to this health disparity dilemma require a new research paradigm for drawing upon Indigenous communities' cultural strengths. In preliminary research, community members report that 'fracking' activities have had a profound negative impact on their entire way of life. To heal historical trauma and counter these negative dynamics, there must be an acknowledgement and understanding of these "colonially generated cultural disruptions. " By understanding the ways in which these external and internal processes occurred and continue to operate, some Indigenous communities are beginning to further understand historical trauma and its consequences as well as identifying their own cultural strengths to overcome or transcend them through community-engaged research approaches. Decolonizing methodologies that use Indigenous-centered approaches can help to engage a community in transformative action.

Culture: An Under-Appreciated Indigenous Asset. Culture is often ignored, devalued, or under-conceptualized in health interventions. However, in Indigenous communities, collective cultural knowledge and community cultural wealth continues to inform and sustain contemporary ways of life Yet, much of this system of Indigenous knowledge has been marginalized, largely underutilized and eroded, and this is particularly true in relation to health research. Movement away from Indigenous cultural practices and decreasing usage of Indigenous language has made indigenous conceptualization of wellbeing at individual, family, and community levels difficult. Increasingly, however, Indigenous communities are working to recover, reclaim, revitalize, and restore their cultural knowledge about wellbeing, including language, traditional economies, and traditional ecological knowledge. They are recognizing to draw on cultural strengths to maintain relationships and partnerships that will be sustainable for future generations. They are using Indigenous-centered approaches and traditional cultural understandings to guide and inform community-based research projects and initiatives. Indigenous communities and researchers are re-centering Indigenous cultural knowledge to structure research with Indigenous communities by finding new ways to transcend the impacts of historical trauma, cultural genocide, environmental degradation, and internalized oppression. Community based participatory research by Indigenous scholars working with Indigenous communities can examine these critical issues while considering strategic ways in planning for and implementing effective transformational changes to address behavioral and mental health disparities that have not been responsive to more traditional approaches.

Theoretical Frameworks and Decolonizing Methodologies for Tribal Health Research. Community Based Participatory Research (CBPR): Research with Indigenous communities has increasingly turned to CBPR approaches to reduce disparities and strengthen wellness . CBPR is not a research method per se, but is an orientation that challenges the traditional roles of researcher and researched to examine their roles of power, participation (who is included and who excluded) and who is leading the knowledge creation agenda; and as such, directly, address the aims of this study by reducing mistrust between the academy and the communities. Tribal Critical Theory: Brayboy's Tribal Critical (Crit) Theory emphasizes how "concepts of culture, knowledge, and power take on new meaning when examined through an Indigenous lens" and the way "tribal philosophies, beliefs, customs, traditions, and visions for the future are central to understanding the lived realities of Indigenous people" significant implications for change at the individual, family, and community level. For example, when research is used as an intervention as embedded within the goals of a research project, the research process allows for community engagement and partnerships to grow in a way that is essential to creating safe spaces for critical community dialogue and praxis with a focus on moving towards healing. Diné-Centered Scientific Research (DCSR) Methodology: DCSR is based on the Hózhóogo Na'aadá evaluation process . The Hózhóogo Naa'adá model was developed by the late Dr. Larry Emerson and Dr. Herbert Benally through a UNM P20 grant titled Our Journey Together. This research methodology allows for the utilization of a Diné-centered research lens to identify, evaluate, and assess life on the Navajo Nation and praxis to resolve these issues using culturally appropriate principles and values like K'é. K'é is the Diné (Navajo) kinship system that honors and recognizes relationships with family, relatives, and others based on the core values of love, respect, reciprocity, and responsibility.

APPROACH. Overview: The proposed study will create a university-community research partnership and increase community member capacity for research in 3 Indigenous communities in New Mexico (NM) using a culture-based lens. The Navajo communities of Counselor, Ojo Encino, and Torreon/StarLake are located in northwestern New Mexico in the easternmost part of the Navajo reservation lands. The overall population of the communities is relatively a younger population with the average household income of under $20,000 and an unemployment average of about 20%. Moreover, these communities much like other Indigenous are experiencing many health disparities. All of these communities experienced a decline in population since the 1990s due to undercounting and/or community members leaving to seek employment in border towns like Farmington. Each community's local governing body or chapter house is part of the Navajo Nation's Eastern agency chapter government system. They have partnered to create a Tri-Chapter alliance to create an equitable system of revenue sharing to address local issues like oil and gas operations and road improvement as well as public safety, education, and community development. All of these communities are located in the Eastern checkerboard area of the Navajo nation consisting primarily Bureau of Land Management (BLM) lands, individual land allotments, Navajo trust lands, and private lands owned by non-Navajos. Many families living in these communities live on allotments that are currently being impacted by oil and gas drilling operations. In January 2018, a grassroots movement focused on the explosive growth of oil and gas activity in the northwest region of the state particularly on the Navajo Nation combined their resources to propose a health study focused on a Health Impact Assessment (HIA) of the three Navajo chapters. Therefore, the investigators will engage community members in critical dialogue about recovering Indigenous knowledge and regenerating Indigeneity, our hypothesis and research design are based on a Tribal Crit theoretical framework that aims to explore the perspectives of community members' understandings of well-being from a Diné centered paradigm using a CBPR approach integrated with a DCSR methodology. The proposed project will develop a Dine conceptualization of well-being with plans to build upon this knowledge through future studies to develop a community profile survey in the hopes of obtaining baseline community health information that can be monitored as oil and gas activities are expected to increase over the next decade. The PI will submit and obtain both UNM and Navajo IRB approvals and all participants will provide signed informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Navajo community member
* Adults over the age of 18) from one of the three Navajo communities
* Local community health service providers and/or tribal employees
* Local tribal leaders and/or educators

Exclusion Criteria:

* Community members who are under 18

Ages: 18 Years to 102 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The main requirement for participation in this study is self-identifying as a Navajo community member (adult or elder over the age of 18) from one of the three Navajo communities. Also emphasized in this study are community tribal and (possibly) non-tribal members who are service providers and/or tribal employees who work with the local community schools, behavioral health or social service organizations..
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2018-03-17 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Developing Community Partnerships | 4 months
  This community based participatory research project was designed as an intervention process to demonstrate an increase in community capacity in doing research using an Indigenous centered approach to engaging with community members in Indigenous contexts by drawing upon their cultural perspectives about partnership, collaboration, trust, reciprocity, and respect. A primary outcome will be the application of a community engagement survey will be used to measure these aspects of developing community partnerships in research especially with Indigenous communities. The community engagement survey tool had 91 items using a likert scale that asked specific questions about how community members were engaged in the process of research.
Defining Community Well-Being | 4 months
  This community based participatory research project was designed as an intervention process to enable the development of a behavioral/mental health framework using key cultural aspects of K'é related to affirming relationships at the familial and community levels. By emphasizing these aspects drawn from local cultural practices and knowledge for community engagement, the study aimed to define community wellbeing with community partners. A primary outcome will be the development of a wellbeing framework for use in future behavioral and mental health research.

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No